CLINICAL TRIAL: NCT02665156
Title: Phase 2 Clinical Trial to Assess Time Efficiency of Intracorporeal Orthotopic Diversion With Robotic Staplers After Robot Assisted Radical Cystectomy
Brief Title: Time Efficiency of Intracorporeal Orthotopic Diversion With Robotic Staplers After Robot Assisted Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Principal Investigator, Giuseppe SImone, Ph.D., Regina Elena Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1034/15
Record Dates: First submitted 2016-01-19; First posted 2016-01-27 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Cystectomy; Robotic Surgical Procedures; Surgical Staplers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robotic Stapled orthotopic neobladder (Experimental): Intracorporeal stapled neobladder using robotic staplers: Partly stapled orthotopic neobladder: robotic staplers applied to create the neobladder neck and to suture the left side of the posterior aspect of neobladder. Right side of the posterior aspect of neobladder and the anterior aspect of the neobladder hand sewn.
  Interventions: Procedure: Intracorporeal stapled neobladder using robotic staplers

INTERVENTIONS:
Procedure: Intracorporeal stapled neobladder using robotic staplers — Robot assisted radical cystecomy. Separate packages extended pelvic lymph node dissection up to aortic bifurcation. Totally intracorporeal orthotopic ileal neobladder with about 45 cm of ileum according to "Vescica Ileal Padovana".

SUMMARY:
Objectives and Specific Aims Time efficiency of robot assisted radical cystectomy (RARC) with totally intracorporeal stapled orthotopic neobladder remains a main drawback of this procedure. According to a recent consensus panel, the benchmark for intracorporeal orthotopic neobladder should be 5 hours in high volume centers .

This prospective single-stage phase 2 trial is designed to assess the time efficiency of using robotic stapler versus the conventional motorized staplers (Linear stapler articulated Endo GIA™, Covidien) in achieving the target outcome (total operative time <5 hr).

Perioperative complications (intraoperative and 30-d postoperative complications according to the Clavien classification system), 30-d/90-d/ 180-d complication and readmission rates, early functional outcomes (time to recovery of urinary continence), 180-d and 360-d neobladder stone formation rates will be analyzed to assess the safety and the cost effectiveness of the procedure.

DETAILED DESCRIPTION:
The primary end point by which the sample size was determined was a total operative time <5hr. In the last 50 cases of our series (data unpublished) this benchmark was obtained in 60% of patients (p0), while we expect to improve the time efficiency of the procedure with the use of robotic staplers maintaining the total operative time of the procedure <5hrs in at least 80% (p1) of cases. According to A'Hern, in order to verify the significance of this hypothesis, the estimated sample size is 33 patients with a power of 80% at a significance level of 5%. The trial will be successful if the total operative time will be <5hrs in at least 25 out of 33 patients.

The population of this study will include 35 patients with muscle invasive bladder cancer without contraindications to orthotopic neobladder. The first two cases will be excluded in order to provide the entire surgical team the minimal skill necessary for a proper and time efficient use of the new surgical device (robotic stapler). The following 33 consecutive cases will be enrolled and the outcomes analyzed. The estimated time to complete the enrollment is 9 months.

ELIGIBILITY:
Inclusion Criteria:

- Pathologically confirmed muscle invasive bladder cancer or recurrent high grade urothelial carcinoma (BCG failures)

Exclusion Criteria:

* All absoulte contraindications to orthotopic neobladder;
* Anesthesiologic contraindications to penumoeperitoneum and steep Trendelenburg position.
* cT4 disease;
* clinical evidence of metastases (cM1) outside the pelvis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Improving time efficiency, achieving a total operative <5 hrs in 80% of cases (28/33) | 1 yr

SECONDARY OUTCOMES:
Perioperative complications | 6 months
  Assessment of perioperative complications 30 days, 90 days and 180 days after surgery
Readmission rate | 6 months
  Incidence of readmission
Neobladder stone formation | 1-yr
  Incidence of neobladder stone formation
Cost analysis | 1-yr

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Simone, Ph.D., Principal Investigator — "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy